CLINICAL TRIAL: NCT04142957
Title: COPD Pal Phase 1: Assessing the Usability and Acceptability of a Self-management App for Chronic Obstructive Pulmonary Disease
Brief Title: COPD Pal Phase 1: A Self-management App in COPD
Status: Completed | Type: Observational
Sponsor: Hywel Dda Health Board (Other)
Collaborators: Welsh Government (Unknown); Bond Digital Health Ltd. (Unknown); Bevan Commission (Unknown)
Responsible Party: Sponsor
Other Study IDs: 270736
Record Dates: First submitted 2019-10-25; First posted 2019-10-29 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: COPD
Keywords: COPD; Self-management; Qualitative; Empowerment; Telehealth
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Empowerment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Focus Groups: The investigators will invite 13-15 participants to attend the focus groups, of which it is expected that 10-12 to attend. Participants will be asked to bring a smart phone. An Informed Consent Form will be signed by the participant and a delegated researcher before the focus groups begin.
  The current generation of COPD Pal will be downloaded onto the participants' own smart phones (see Appendix 1 for current screenshots of app), participants will then be explained the purpose of the app, and asked to interact with it for 15-60 minutes, as required.
  A semi-structured focus group will then be conducted with the participants to facilitate conversation and discussion regarding COPD Pal. Once introductions have been completed, questions will be asked relating to the usability and acceptability of COPD Pal (see the Interview Schedule, Appendix 2). The focus group will last 30-60 minutes, as required.
  Interventions: Other: COPD Pal

INTERVENTIONS:
Other: COPD Pal — 'COPD Pal' aims to allow people with COPD to track and manage their condition. It enables patients to log symptoms (e.g. COPD assessment Test), wellness (e.g. quality of life such as EQ-5D), and medications, to help them become more engaged in their own care.

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a widespread condition which causes a poorer health status, reduced exercise, and lung function impairment. COPD exacerbations are a sustained worsening of symptoms beyond day-to-day variation and are responsible for one in eight hospital emergency admissions. Although extensive users of healthcare, people with COPD are primarily responsible for their condition 99% of the time and self-management has been highlighted as a crucial component for COPD care. To enable greater awareness of changing symptoms, a self-management app (COPD Pal) will be created by Bond Digital Health Ltd (BDH) to enable people with COPD to input information pertinent to their condition. The aim of COPD Pal, which is akin to a paper diary, is to empower patients to take more control of their disease and allow them to provide healthcare professionals with accurate, personalised data during clinic consultations.

This project aims to assess the usability and acceptability of COPD Pal using qualitative methodology (phase 1). It is proposed that 13-15 people with COPD will be invited to attend a focus group and be given COPD Pal (V1) with which to interact. Semi-structured questions will then be asked to facilitate conversation regarding their initial experiences of using COPD Pal. Focus groups will be audio-recorded, transcribed, and a Thematic Analysis conducted. Thematic themes will be provided to BDH, the creators of COPD Pal, with which to develop the app further (V2). Thematic themes will be provided to participants to confirm accuracy and ensure methodological rigour. A final report will be provided to both research participants and to BDH.

Findings from this research will inform the second phase feasibility study of V2 of COPD Pal.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is a global problem, with 210 million sufferers and 3 million deaths annually. It is predicted to become the third most common cause of death worldwide by 2030. There are 1.2 million people with known COPD in the UK, but this is likely to be an underestimate. People with COPD have daily symptoms, a poorer health status, reduced exercise capacity, and impairment in lung function. A sustained worsening of symptoms above day-to-day variation, in response to infection or pollution, is termed an acute exacerbation. Exacerbations of COPD are the second most common cause of emergency admission to hospital in the UK, being responsible for one in eight (130,000) of the total, as well as 1 million bed days and an annual National Health Service (NHS) expenditure of over £500M in 2015.

Despite people with the condition being extensive users of the NHS, approximately only 1% of their time is spent with healthcare professionals. The rest of the time, people with COPD are encouraged to self-manage their condition; where, such behaviours include regular exercise, taking prescribed medication, being aware of symptoms, and attending healthcare appointments. Supporting self-management behaviours has been highlighted as crucial for the care of people with COPD. Despite the positive relationship between self-management and health outcomes, these behaviours are seldom conducted and adherence to medication is historically low.

To enable greater awareness of the change of his symptoms (i.e. better self-management), Ian Bond - who lives with COPD - created a simple diary which allowed him to identify when he was likely to have an exacerbation and thus take preventative action. Creating Bond Digital Health Ltd. (BDH; Cardiff, UK; https://bondhealth.co.uk/) he transformed this paper tool into a basic electronic diary. This quickly evolved into the development of an easy-to-use smart phone app. 'COPD Pal' aims to allow people with COPD to track and manage their condition. It enables patients to log symptoms (e.g. COPD assessment Test), wellness (e.g. quality of life such as EQ-5D), and medications, to help them become more engaged in their own care.

Showing their digital health data to a healthcare professional, during the consultation (by the patient), can guide communication, and empower the patient to lead their clinic appointment, and to become more positively involved in their own care. It should also help any healthcare professional in looking at trends and changes (or consistencies) from baseline health status which are unique for that patient. It is akin to a patient bringing a paper diary to show their healthcare professional the day-to-day variation in their chronic disease.

By improving self-management, illness understanding, and confidence in people with COPD, the app allows greater locus of control and hopefully will lead to reduced GP contacts, number and length of hospitalisations, and present real and immediate cost-savings to the NHS.

Welsh Government have funded (Efficiency through Technology Programme (ETTP), Social Research Number: 51/2017) a collaborative project between BDH and Hywel Dda University Health Board (HDUHB). BDH and their specialist software engineers are developing the prototype, working app. HDUHB have been funded (£16,000) to conduct a quantitative clinical trial and patient focus groups in the later design phases of the app to investigate suitability and usability, and test early feasibility in a real-world setting. It is hoped that such a study could also help improve these aspects for future versions of COPD Pal.

This project describes the Clinical Phase 1, focus groups and aims to answer the research question: 'how do people with COPD experience the usability and acceptability of the COPD Pal app?'

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent.
* Clinical diagnosis of COPD as defined by GOLD (Vogelmeier, et al., 2018; https://goldcopd.org/wp-content/uploads/2018/11/GOLD-2019-v1.7-FINAL-14Nov2018-WMS.pdf), i.e. greater than 40 years old, ≥ 10 pack years smoking history, post-bronchodilator FEV1/FVC ratio of 0.7, with FEV1 less than 80% predicted.
* Owns, or has access to, a smart phone.

Exclusion Criteria:

* Unwilling or unable to provide written informed consent.
* Cognitive, visual, or hearing impairment which would affect communication in a group-setting or ability to see and use a smart phone.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 15 people meeting the criteria above
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Thematic Themes | 2 hours
  The Investigators will conduct focus groups to obtain qualitative data (i.e. no scale will be used)

CONTACTS AND LOCATIONS:
Overall Officials: Liam Knox, Principal Investigator — Hywel Dda University Health Board
Locations (1):
- Prince Philip Hospital, Llanelli, Carmarthenshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided